CLINICAL TRIAL: NCT04792853
Title: Tablet-based Cognitive Behavioral Intervention: Comparison of Group vs. Individual CBT Education
Brief Title: Tablet-based Cognitive Behavioral Intervention for Older Adults With Arthritis Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Jeungok Choi, Associate professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2130
Record Dates: First submitted 2021-03-07; First posted 2021-03-11 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Arthritis; Fatigue
Keywords: arthritis; fatigue; cognitive behavioral therapy; group education; older adults; tablet; simple walking
MeSH Terms: conditions — Arthritis; Fatigue

STUDY DESIGN:
Intervention Model Description: The study uses an experimental pre- and post-test repeated measures design. Those satisfying the inclusion and exclusion criteria are randomly assigned to the intervention (Tab-G, n=20) or comparison group (n=20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tab-G (tablet-based group CBT education) (Experimental): Tab-G participants will receive 4 weekly CBT(cognitive behavioral therapy)-based group learning sessions to encourage a simple walking activity through videoconferencing meetings in a group of 5 members. The educational materials emphasize shared goal setting and mutual reinforcement.
  Interventions: Behavioral: Tab-G
- Usual care group (No Intervention): A usual care group will receive general arthritis management education. Participant are instructed to maintain usual activity during the study period.

INTERVENTIONS:
Behavioral: Tab-G — Participants receive a tablet preloaded with Tab-G application and an accelerometer.
  Other Names: tablet-based group CBT education
  Arms: Tab-G (tablet-based group CBT education)

SUMMARY:
The purpose of this project is to pilot test a long-term effect of Tab-G (tablet-based cognitive behavioral group education intervention). The investigators will evaluate the effect of Tab-G, relative to usual care group, on (a) daily steps, (b) fatigue level, (c) self-efficacy and (d) quality of life.

Tab-G participants will receive 4 weekly CBT-based group education focusing on shared goal setting and mutual reinforcement in a group with 5 members. The outcomes will be measured baseline, week 4 (intervention completion) and week 8 (follow-up). The investigators hypothesize that older adults receiving Tab-G will have greater improvements on outcomes compared to those receiving usual care at week 4, the intervention completion and at week 8 follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of osteoarthritis or rheumatoid arthritis;
2. presence of greater than minimal fatigue scoring ≥13 (T-score>55) on the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v1.0-Fatigue 6a; and
3. having Wi-Fi at home

Exclusion Criteria:

1. currently engaging in regular exercise;
2. non-ambulatory or presence of a condition that would limit the ability to walk (e.g., foot deformity, lower extremity joint surgery in past 6 months, stroke, severe chronic obstructive pulmonary disease, etc.); and
3. delirium, dementia, or any conditions indicating deteriorating cognitive status as determined by the Mini-Cog.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
daily steps | 24 hours
  daily step counts measured by an accelerometer
BRICS NINR PROMIS Fatigue Short Form 6a | past 1 week
  self-reported fatigue scale measuring both the experience of fatigue and the interference of fatigue on daily activities. Scores can range from 6 to 30, with higher scores indicating greater fatigue.
Self-Efficacy for Managing Chronic Disease 6-Item Scale | 24 hours
  self-reported self-efficacy scale. Scores can range from 6 to 60, with higher scores indicating higher self-efficacy.
Quality of Life-Rheumatoid Arthritis Scale | past 4 weeks
  self-reported perception of quality of life. Scores can range from 8 to 80 with higher scores indicating greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jeungok Choi, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States